CLINICAL TRIAL: NCT05616377
Title: Survival Benefit of Combination of Local Therapy and Target Therapy for Brain Metastases With EGFR Mutation: A Multicenter Retrospective Study
Brief Title: Combination of Local Therapy and Target Therapy for Brain Metastases With EGFR Mutation
Acronym: CLTBME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yonggao Mou, Department of Neurosurgery, Sun Yat-sen University
Other Study IDs: EGFR+BM
Record Dates: First submitted 2022-11-08; First posted 2022-11-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative; Radiotherapy; Lead

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- target therapy + local therapy group vs target therapy alone group
  Interventions: Other: Surgery or Radiotherapy
- local therapy before target therapy group vs local therapy after target therapy group
  Interventions: Other: before or after target therapy

INTERVENTIONS:
Other: Surgery or Radiotherapy — Participants who underwent target therapy and surgery or radiotherapy were divided into target therapy + local therapy group. Participants who underwent target therapy alone were divided into target therapy alone group
  Groups: target therapy + local therapy group vs target therapy alone group
Other: before or after target therapy — Participants who underwent surgery or radiotherapy before target therapy were divided into local therapy before target therapy group. Participants who underwent surgery or radiotherapy after target therapy were divided into local therapy after target therapy group.
  Groups: local therapy before target therapy group vs local therapy after target therapy group

SUMMARY:
The goal of this observational study is to learn about the survival benefit of local therapy combination with target therapy in lung cancer brain metastases with EGFR mutation. The main questions it aims to answer are:

* Is local therapy performed before or after target therapy would provide survival benefit ?
* What kind of local therapy combining with target therapy would provide survival benefit, neurosurgical resection or radiotherapy?

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of pathological diagnosis of primary tumor.
2. Brain metastases confirmed by enhanced magnetic resonance imaging.
3. Gene test indicated that EGFR mutation.
4. Complete clinical information.

Exclusion Criteria:

1. If surgical treatment is accepted, the surgical treatment is not tumor resection, but ventricle puncture, biopsy and other non-tumor reducing surgery.
2. Patients with 2 or more types of tumors.
3. Incomplete clinical information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital clients from Sun Yat-sen University Cancer Center, Guangxi Medical University Cancer Hospital, The People's Hospital Of Guangxi Zhuang Autonomous Region, and the First Affiliated Hospital of Guangxi Medical University will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-11-20 (Estimated); Primary Completion 2023-08-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
OS | From date of first follow-up until the date of documented death from any cause, assessed up to 120 months
  Overall survival

SECONDARY OUTCOMES:
PFS | From date of first follow-up until the date of first documented progression, assessed up to 120 months
  Progression-free survival

IPD SHARING:
Plan to Share IPD: Undecided